CLINICAL TRIAL: NCT00638924
Title: Analysis of Physiologic Variables in Healthy Women in Shuttle Walk Test
Brief Title: Physiologic Variables in Healthy Women in Shuttle Walk Test
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Juliana Gomes Z|abatiero, Student, University of Campinas, Brazil
Other Study IDs: 200802
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: healthy sedentary women

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exercise Capacity: Individuals from the female gender; age range of 20 to 30 years old; considered healthy (i.e. with no diagnosed health condition; considered sedentary (i.e. performing less than 150 minutes of moderate intensity physical activity per week); will be asked to volunteer in the research and perform a exercise capacity test.
  Interventions: Other: Shuttle walk test

INTERVENTIONS:
Other: Shuttle walk test — the test requires patients to walk at a gradually increasing speed, up and down a 10 m course identified by two marker cones, until they reach a symptom limited maximum. The walking speed was externally paced and controlled by a series of beeps played on a compact disk.
  Other Names: Shuttle Walking Test; Exercise Capacity Test

SUMMARY:
To analyze the alterations of physiologic variables in healthy sedentary women in the Shuttle Walk Test, verify the distance reached and interruption causes of the test.

DETAILED DESCRIPTION:
The Shuttle Walk Test requires patients to walk at a gradually increasing speed, up and down a 10 meter corridor identified by two marker cones, until they reach a symptom limited maximum. The walking speed was externally paced and controlled by a series of beeps played on a compact disk.

ELIGIBILITY:
1. Inclusion criteria:

   1. female gender;
   2. sedentary;
   3. aged 20 to 30 years.
2. Exclusion criteria:

   1. pregnancy;
   2. enrolment in any regular physical activity program;
   3. diagnosed health conditions.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women, between 20 and 30 years old, healthy and sedentary
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivete Alonso Saad, dr, Study Chair — University of Campinas, Brazil
Locations (1):
- State University of Campinas, Campinas, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Inactive Woman: 40 women, 20 to 30 years old, healthy and sedentary
Period: Overall Study
Arm/Group | Inactive Woman
Started | 40
2 Months | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Inactive Woman
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 40

OUTCOME MEASURES:

1. Secondary Outcome: Heart Rate
Description: Heart rate at baseline
Time Frame: baseline
Population: 20 to 30 years old, healthy and sedentary
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Inactive Woman
Number analyzed (Participants) | 40
bpm | 83.8 (14.4)

2. Primary Outcome: Shuttle Walk Test Distance
Description: The distance achieved in the test in meters
Time Frame: baseline
Population: 20 to 30 years old, healthy and sedentary
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Inactive Woman
Number analyzed (Participants) | 40
m | 812 (165)

ADVERSE EVENTS:
Arm/Group | Inactive Woman
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Small number of subjects, only females were analyzed making generalization impossible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes